CLINICAL TRIAL: NCT05122650
Title: A Phase 2b, 12-week, Double-blind, Placebo-controlled, Randomized, Parallel Group, Multicenter Study of the Safety and Efficacy of JZP385 in the Treatment of Adults With Moderate to Severe Essential Tremor
Brief Title: A Study To Assess the Safety and Efficacy of JZP385 in the Treatment of Adults With Moderate to Severe Essential Tremor (ET)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JZP385-201; 2020-002463-61 (EudraCT Number)
Record Dates: First submitted 2021-11-02; First posted 2021-11-17 (Actual); Results first posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Essential Tremor
Keywords: JZP385; T-type calcium channels; Movement disorder; Tremor; Moderate to severe essential tremor
MeSH Terms: conditions — Essential Tremor; Movement Disorders; Tremor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 10 milligram (mg) JZP385 (Experimental): Participants will initially receive 5 mg/day from Day 1 through Day 7, and 10 mg/day starting on Day 8.
  Interventions: Drug: JZP385
- 20 mg JZP385 (Experimental): Participants will initially receive 5 mg/day from Day 1 through Day 7, 10 mg/day from Day 8 through Day 14, and 20 mg/day starting on Day 15.
  Interventions: Drug: JZP385
- 30 mg JZP385 (Experimental): Participants will initially receive 5 mg/day from Day 1 through Day 7, 10 mg/day from Day 8 through Day 14, 20 mg/day from Day 15 through Day 21, and 30 mg/day starting on Day 22.
  Interventions: Drug: JZP385
- Placebo (Placebo Comparator): Participants will receive placebo from Day 1.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: JZP385 — JZP385 capsules will be administered orally (PO) once daily in the morning on an empty stomach for 12 weeks.
  Arms: 10 milligram (mg) JZP385; 20 mg JZP385; 30 mg JZP385
Other: Placebo — Placebo capsules will be administered orally (PO) once daily in the morning on an empty stomach for 12 weeks.
  Arms: Placebo

SUMMARY:
This is a 12-week, double-blind, placebo-controlled, randomized, parallel-group, multicenter study of the safety and efficacy of JZP385 in the treatment of adult participants with moderate to severe ET.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be 18 to 80 years of age inclusive, at the time of signing the informed consent.
2. Participants who are diagnosed with ET (including ET plus) according to the MDS Consensus Statement on the Classification of Tremors from the Task Force on Tremor of the International Parkinson's and Movement Disorder Society.
3. Participants have moderate to severe disability associated with tremor as determined by a score of ≥ 22 on the TETRAS-ADL subscale and a CGI-S rating of at least moderate for participants' ability to function.
4. Sex and Contraceptive/Barrier Requirements

   During the study intervention and for at least 30 days after the last dose of study intervention male participants must refrain from donating sperm. Non-abstinent males must agree to use a male condom in combination with female partner use of a highly effective contraceptive method with a failure rate of < 1% per year. All male participants must agree to use a male condom when engaging in any activity that allows for passage of ejaculate to another person.

   Female participants must not be pregnant or breastfeeding, are either women of non-childbearing potential (WONCBP), or are women of childbearing potential (WOCBP) using a highly effective contraceptive method with a failure rate of < 1% during the study intervention period and for at least 30 days after the last dose of study intervention. Male partners of WOCBP are required to use barrier protection, eg, condoms, from the first dose of study intervention until 30 days after the last dose of study intervention.

   A WOCBP must have a negative highly sensitive serum pregnancy test at Screening Visit 1 and negative urine pregnancy tests (unless serum is required by local regulations) at the Screening Visit 2 (if applicable) and at the Baseline Visit

   - If a urine test cannot be confirmed as negative (eg, an ambiguous result), a serum pregnancy test is required. In such cases, the participant must be excluded from participation if the serum pregnancy result is positive.
5. Prior/Concomitant Antitremor Medications

If currently treated with antitremor medications, potential participants must be on a stable dosage for at least 6 weeks prior to Screening and must not anticipate making any changes to their antitremor medication for the duration of the study. Note: Treatment with some antitremor medications (eg, primidone) is not allowed in accordance with other exclusion criteria.

Exclusion Criteria:

1. Known history or current evidence of other medical or neurological conditions that may cause or explain the participant's tremor.
2. Has evidence at Screening of severe cognitive impairment as defined by a Montreal Cognitive Assessment (MoCA; score < 20) or has cognitive impairment that in the opinion of the investigator would prevent completion of study procedures (including the ability to accurately self-report on study questionnaires) or the ability to provide informed consent.
3. Current suicidal risk as determined from history, by presence of active suicidal ideation as indicated by positive response to item 4 or 5 on the C-SSRS (within the past 24 months), or any history of suicide attempt; current or past (within 1 year) major depressive episode according to DSM-5 criteria.
4. History (within past 2 years at screening) or presence of a diagnosed substance use disorder (including alcohol, tobacco, and cannabis) according to DSM-5 criteria, known drug dependence, or seeking treatment for alcohol or substance abuse related disorder.
5. Prior magnetic resonance (MR)-guided focused ultrasound thalamotomy, surgical intervention (eg, deep brain stimulation, ablative thalamotomy, gamma knife thalamotomy), or inability to refrain from using a device for treatment of tremor for the duration of the treatment period.
6. Botulinum toxin injection for the treatment of upper limb tremor in the 6 months before screening or planned use at any time during the study.
7. Treatment with any medication that could produce tremor taken within 2 weeks or 5 half-lives (whichever is longer) before screening or anticipated use at any time during participation in the study.
8. Use of prescription of nonprescription drugs or other products known to be inducers of CYP3A4 that are known to decrease AUC by > 30% (eg, primidone) and which cannot be discontinued at least 4 weeks before Baseline or planned use at any time during the study.
9. Use of prescription or nonprescription drugs, or other products (eg, grapefruit, grapefruit juice, or Seville oranges) known to be strong or moderate inhibitors of CYP3A4, that cannot be discontinued 2 weeks or 5 half-lives, whichever is longer, before Baseline or planned use at any time during the study.
10. Use of proton pump inhibitors that cannot be discontinued at least 2 weeks before Baseline, or planned use at any time during the study. Occasional use of antacids or histamine-2 receptor antagonists will be permitted, but antacids should be taken at least 4 hours before or after study intervention; and histamine-2 receptor antagonists should be taken at least 4 hours after and at least 12 hours before study intervention.
11. Inability to refrain from use of medication/substance(s) that might produce tremor or interfere with the evaluation of tremor on study visit days prior to discharge such as, but not limited to, stimulant decongestants, beta-agonist bronchodilators, and alcohol.
12. Regular use of more than 3 units of alcohol per day.
13. Regular consumption of caffeine > 400 mg/day or > 4 cups of coffee per day

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (73):
- United States (41):
  - The University Of Alabama At Birmingham (Uab), Birmingham, Alabama
  - St. Joseph's Hospital and Medical Center (SJHMC) - Barrow Neurological Institute (BNI) - The Gregory W. Fulton ALS and Neuromuscular Disease Center, Phoenix, Arizona
  - Arizona Neuroscience Research, LLC, Phoenix, Arizona
  - Imaging Endpoints II, LLC, Scottsdale, Arizona
  - Movement Disorders Center of Arizona, Scottsdale, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - Pillar Clinical Research, LLC, Bentonville, Arkansas
  - Woodland Research Northwest, LLC, Rogers, Arkansas
  - The Parkinson's and Movement Disorder Institute, Fountain Valley, California
  - Keck School of Medicine USC - Healthcare Consultation Center 2 (HCCII), Los Angeles, California
  - SC3 Research - Beverly, Los Angeles, California
  - SC3 Research Pasadena, Pasadena, California
  - Neurology of Central Florida Research Center, Altamonte Springs, Florida
  - JEM Research Institute, Atlantis, Florida
  - Parkinson's Disease And Movement Disorder Center Of Boca Raton, Boca Raton, Florida
  - Innovative Research Of West Florida, Inc., Clearwater, Florida
  - Infinity Clinical Research, Llc, Hollywood, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Homestead Associates in Research, Inc., Miami, Florida
  - USF Carol and Frank Morsani Center for Advanced Healthcare, Tampa, Florida
  - University of South Florida Parkinson's Disease and Movement Disorders Center, Tampa, Florida
  - Neurotrials Research, Inc., Atlanta, Georgia
  - Brain Health Center, Emory University, Atlanta, Georgia
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - Northwestern University - Feinberg School of Medicine - ParkinsonÃÂ¿s Disease and Movement Disorders Center, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Louisville, Movement Disorder Clinic, Louisville, Kentucky
  - QUEST Research Institute, Farmington Hills, Michigan
  - University Nebraska Medical Center, Omaha, Nebraska
  - Dent Neurological Institute, Amherst, New York
  - South Shore Neurology Associates, Inc., Patchogue, New York
  - University of Rochester Medical Center, Rochester, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Duke University Health System, Durham, North Carolina
  - American Clinical Research Institute LLC, Beavercreek, Ohio
  - NeuroScience Research Center, Canton, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Houston Methodist Hospital - Movement Disorders Clinic, Houston, Texas
  - Booth Gardner Parkinson's Care Center, Kirkland, Washington
  - Vaught Neurological Services, PLLC, Crab Orchard, West Virginia
- Germany (9):
  - Universitaetsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Velocity Clinical Research Germany GmbH, Wiesbaden, Hesse
  - Zentrum for klinische Forschung Dr. med. Irma Schoell, Bad Homburg
  - Pharmakologisches Studienzentrum Chemnitz, Chemnitz
  - University Hospital Duesseldorf, Düsseldorf
  - Klinik Haag i. OB, Haag
  - CRC Core Facility Medizinische Hochschule Hannover (MHH), Hanover
  - DKD HELIOS Klinik Wiesbaden, Wiesbaden
  - Klinikum der Julius-Maximilians-Universitaet Wuerzburg, Würzburg
- Poland (14):
  - Neuro-Care Sp. Z.o.o. sp. Komandytowa, Katowice, Silesian Voivodeship
  - Medicover Integrated Clinical Services (MICS) Centrum Medyczne Bydgoszcz, Bydgoszcz
  - NZOZ Wielospecjalistyczna Poradnia Lekarska Synapsis, Katowice
  - Centrum Medyczne Plejady, Krakow
  - Specjalistyczne Gabinety Sp. z o.o, Krakow
  - Landa Specjalistyczne Gabinety Lekarskie, Krakow
  - Krakowska Akademia Neurologii Sp. z o.o, Krakow
  - Linden Centrum Medyczne, Krakow
  - Niepubliczny Zaklad Opieki Zdrowotnej (NZOZ) Neuromed M. i M. Nastaj Spolka Partnerska( Sp.P.), Lublin
  - Centrum Zdrowia I Urody Maxxmed, Lublin
  - Neurologiczny NZOZ Centrum Leczenia SM Osrodek Badan Klinicznych im. dr n. med. Hanki Hertmanowskiej, Plewiska
  - Rivermed Sp z o.o, Poznan
  - ETG Neuroscience, Warsaw
  - MD Clinic Praga Spolka z o. o., Warsaw
- Spain (9):
  - Hospital Universitario Virgen Macarena-merge, Seville, Andalusia
  - CAE Oroitu (Centro de Atencion Especializada), Getxo, Vizcaya
  - Hospital de Cruces, Barakaldo
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Policlinica Gipuzkoa, Donostia / San Sebastian
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Puerta de Hierro de Majadahonda, Majadahonda

IPD SHARING:
Plan to Share IPD: Yes
In accordance with ICMJE requirements, Jazz Pharmaceuticals may provide qualified external researchers access to individual participant data (IPD) and clinical trial data that underlie the results of this trial upon request. Qualified researchers can submit a request on https://www.jazzpharma.com/science/clinical-trial-data-sharing/ as outlined. Jazz Pharmaceuticals reserves the right not to consider a request. For inquiries about Jazz's data sharing policy contact clinicaldatasharing@jazzpharma.com.
URL: https://www.jazzpharma.com/science/clinical-trial-data-sharing

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 420 participants were randomized to treatment. These 420 participants are included in the Intent to Treat Analysis set (ITT). Of those 420 participants, only 416 received at least 1 dose of study intervention. Four participants did not receive any treatment. These 416 participants are included in the Safet Analysis Set
Period: Overall Study
Arm/Group | Placebo | 10 Milligram (mg) JZP385 | 20 mg JZP385 | 30 mg JZP385
Started | 104 | 105 | 104 | 107
Completed | 91 | 78 | 81 | 78
Not Completed | 13 | 27 | 23 | 29
Not completed — Adverse Event | 4 | 16 | 11 | 12
Not completed — Lack of Efficacy | 0 | 1 | 1 | 2
Not completed — Lost to Follow-up | 1 | 1 | 3 | 0
Not completed — Non-compliance with study intervention | 0 | 0 | 0 | 2
Not completed — Protocol Violation | 0 | 1 | 0 | 1
Not completed — Randomized by mistake | 0 | 0 | 3 | 2
Not completed — Sponsor request | 0 | 1 | 1 | 2
Not completed — Withdrawal by Subject | 3 | 7 | 4 | 8
Not completed — Other | 5 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 10 Milligram (mg) JZP385 | 20 mg JZP385 | 30 mg JZP385 | Total
Number analyzed (Participants) | 104 | 105 | 104 | 107 | 420
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 43 | 51 | 45 | 48 | 187
  >=65 years | 61 | 54 | 59 | 59 | 233
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 37 | 33 | 49 | 160
  Male | 63 | 68 | 71 | 58 | 260
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 10 | 9 | 11 | 41
  Not Hispanic or Latino | 93 | 95 | 95 | 96 | 379
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 4 | 4 | 8
  White | 98 | 96 | 93 | 92 | 379
  More than one race | 0 | 1 | 1 | 2 | 4
  Unknown or Not Reported | 5 | 7 | 6 | 9 | 27

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 on the TETRAS Composite Outcome Score as Summarized by Each Dose of JZP385 and Placebo
Description: The TETRAS composite outcome score is the sum of modified items 1 - 11 of the TETRAS-ADL subscale and modified items 6 - 7 of the TETRAS-PS. The TETRAS-ADL subscale is a patient-rated scale administered by a trained interviewer that assesses the impact of tremor on day-to-day functioning, such as eating, drinking, dressing, and other fine motor skills. The TETRAS-PS is a clinical rating scale that quantifies tremor in the head, face voice, limbs and trunk. Items 6 (drawing an Archimedes spiral using left and right hands) and 7 (handwriting) of the TETRAS-PS evaluate the impact of upper limb tremor on performance. Each item from the modified subscales ranges from 0 - 3, with 0 representing normal or slightly abnormal and 3 representing severely abnormal. The sum of the 14 items provides the TETRAS composite outcome score, which ranges from 0 - 42, with higher scores representing more severe ET.
Time Frame: Change from baseline to week 12
Population: The primary outcome was assessed in participants in the Intent to Treat (ITT) analysis population set that completed the baseline and week 12 TETRAS assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | 10 Milligram (mg) JZP385 | 20 mg JZP385 | 30 mg JZP385
Number analyzed (Participants) | 94 | 79 | 82 | 78
score on a scale | -6.3 (6.22) | -5.8 (6.85) | -6.7 (6.88) | -7.5 (7.31)

2. Secondary Outcome: Percentage of Participants Who Improved (≥ 1-Point Improvement) From Baseline to Week 12 on the Clinical Global Impression- Severity Scale (CGI-S)
Description: The CGI-S is a 5-point Likert-type rating scale that a qualified medical personnel (ie, a clinician)will use to rate the severity of the participants' ability to function due to their ET. The responses to this scale range from 1 (no limitations) to 5 (severe).
Time Frame: Change from baseline to week 12
Population: Inferential analysis results were based on multiple imputations (impute missing values) on all study population
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | 10 Milligram (mg) JZP385 | 20 mg JZP385 | 30 mg JZP385
Number analyzed (Participants) | 104 | 105 | 104 | 107
Percentage of participants | 50.0 | 49.8 | 55.7 | 62.8

3. Secondary Outcome: Proportion of Participants Reported as Much Improved on the Clinical Global Impression of Change (CGI-C) at Week 12
Description: The CGI-C is a 5-point Likert-type rating scale that a qualified medical personnel (ie, a clinician) will use to rate the change in severity of the participants' ability to function due to their ET since baseline. The responses to this scale range from 1 (Much improved) to 5 (Much worse).
Time Frame: Week 12
Population: The outcome was assessed in participants in the Intent to Treat (ITT) analysis population set that completed the baseline and week 12 CGI-C assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 10 Milligram (mg) JZP385 | 20 mg JZP385 | 30 mg JZP385
Number analyzed (Participants) | 94 | 79 | 82 | 79
Participants | 22 | 18 | 19 | 30

4. Secondary Outcome: Proportion of Participants Reported as Much Improved on the Patient Global Impression of Change (PGI-C) at Week 12
Description: The PGI-C is a 5-point Likert-type rating scale that participants use to rate the change in severity of their ability to function due to ET since baseline. The responses to this scale range from 1 (Much improved) to 5 (Much worse).
Time Frame: Change from baseline to week 12
Population: The outcome was assessed in participants in the Intent to Treat (ITT) analysis population set that completed the baseline and week 12 PGI-C assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 10 Milligram (mg) JZP385 | 20 mg JZP385 | 30 mg JZP385
Number analyzed (Participants) | 94 | 79 | 82 | 79
Participants | 16 | 11 | 20 | 32

5. Secondary Outcome: Change From Baseline to Week 12 on the TETRAS-ADL Subscale as Summarized by Each Dose of JZP385 and Placebo
Description: The TETRAS-ADL subscale is a patient-rated scale of the impact of tremor on day-to-day functioning administered by a trained interviewer. The TETRAS-ADL subscale directly measures how a patient functions by assessing activities impacted by tremor, such as eating and drinking, dressing and personal hygiene, carrying items and fine motor skills. The TETRAS-ADL has 12 items, and each item is rated on a 0 (normal) to 4 (severe) scale with a total score ranging from 0 to 48. A higher score represents more severe ET.
Time Frame: Change from baseline to week 12
Population: The outcome was assessed in participants in the Intent to Treat (ITT) analysis population set that completed the baseline and week 12 TETRAS-ADL assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | 10 Milligram (mg) JZP385 | 20 mg JZP385 | 30 mg JZP385
Number analyzed (Participants) | 94 | 79 | 82 | 79
score on a scale | -6.4 (6.40) | -6.3 (7.55) | -7.1 (7.88) | -8.7 (8.49)

6. Secondary Outcome: Change From Baseline to Week 12 on the TETRAS-PS Subscale as Summarized by Each Dose of JZP385 and Placebo
Description: The TETRAS-PS is a clinical rating scale performed by a blinded rater that quantifies tremor in the head, face, voice, limbs, and trunk. Each item will be rated on a scale of 0 (normal) to 4 (severe). The sum of the individual scores provides the overall score, ranging from 0 to 64, with higher scores representing more severe ET.
Time Frame: Change from baseline to week 12
Population: The outcome was assessed in participants in the Intent to Treat (ITT) analysis population set that completed the baseline and week 12 TETRAS-PS subscale assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | 10 Milligram (mg) JZP385 | 20 mg JZP385 | 30 mg JZP385
Number analyzed (Participants) | 94 | 79 | 82 | 78
score on a scale | -5.4 (5.73) | -5.3 (6.57) | -5.1 (6.15) | -5.5 (6.27)

7. Secondary Outcome: Change From Baseline to Week 12 on the Upper Limb Score (Item 4) of the TETRAS-PS as Summarized by Each Dose of JZP385 and Placebo
Description: Item 4 of the TETRAS-PS measures upper limb tremor, and includes 3 maneuvers for each arm that assess postural and kinetic tremor. Each item is rated on a scale of 0 (normal) to 4 (severe) in 0.5-point increments. The total score is the sum of each of the 6 items and ranges from 0 to 24, with higher scores representing more severe ET. The TETRAS-PS is performed by a blinded rater.
Time Frame: Change from baseline to week 12
Population: The outcome was assessed in participants in the Intent to Treat (ITT) analysis population set that completed the baseline and week 12 Upper limb score on the TETRAS-PS assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | 10 Milligram (mg) JZP385 | 20 mg JZP385 | 30 mg JZP385
Number analyzed (Participants) | 94 | 79 | 82 | 78
score on a scale | -2.3 (2.68) | -2.4 (2.78) | -2.0 (2.61) | -2.4 (2.81)

8. Secondary Outcome: Change From Baseline to Week 12 on the TETRAS Total Score, as Summarized by Each Dose of JZP385 and Placebo.
Description: The TETRAS total score is the sum of the scores of the full TETRAS-ADL and TETRAS-PS subscales. Each item is rated on a 0 (normal) to 4 (severe) scale, and total scores range from 0 to 112, with higher scores representing more severe ET. The TETRAS-PS is performed by a blinded rater.
Time Frame: Change from baseline to week 12
Population: The outcome was assessed in participants in the Intent to Treat (ITT) analysis population set that completed the baseline and week 12 TETRAS Total assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | 10 Milligram (mg) JZP385 | 20 mg JZP385 | 30 mg JZP385
Number analyzed (Participants) | 94 | 79 | 82 | 78
score on a scale | -11.8 (10.18) | -11.6 (11.54) | -12.3 (11.95) | -14.4 (12.20)

9. Secondary Outcome: Change From Baseline to Week 12 on the Quality of Life in Essential Tremor Questionnaire (QUEST) as Summarized by Each Dose of JZP385 and Placebo
Description: The Quality of Life in Essential Tremor Questionnaire (QUEST) was developed to specifically assess the impact of ET on health-related quality of life. The QUEST is a 30-item questionnaire comprising 5 subscales (physical, psychosocial, communication, hobbies/leisure, and work/finance). Each item is rated by frequency on a scale from 0 (never) to 4 (always). Each dimension had been standardized to a range of 0 to 100 with higher scores indicating greater dissatisfaction or disability due to ET.
Time Frame: Change from baseline to week 12
Population: The outcome was assessed in participants in the Intent to Treat (ITT) analysis population set that completed the baseline and week 12 QUEST assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | 10 Milligram (mg) JZP385 | 20 mg JZP385 | 30 mg JZP385
Number analyzed (Participants) | 99 | 100 | 95 | 98
score on a scale
  Communication Subscale Total Score | -5.5 (15.35) | -3.3 (15.62) | -3.5 (14.67) | -7.8 (16.18)
  Work and Finance Subscale Total Score | -5.8 (16.44) | 1.0 (17.26) | -6.1 (15.61) | -6.7 (15.11)
  Hobbies and Leisure Subscale Total Score | -1.1 (29.35) | -8.9 (31.66) | -3.5 (36.50) | -10.2 (33.81)
  Physical Subscale Total Score | -11.0 (17.65) | -5.1 (17.60) | -10.1 (16.85) | -13.4 (20.24)
  Psychosocial Subscale Total Score | -6.8 (14.93) | -2.9 (16.57) | -6.1 (15.79) | -6.2 (15.40)

10. Secondary Outcome: Change From Baseline to Week 12 on the Essential Tremor Embarrassment Assessment (ETEA) Score A as Summarized by Each Dose of JZP385 and Placebo
Description: The Essential Tremor Embarrassment Assessment (ETEA) is a participant-rated questionnaire administered by a health care provider or researcher that contains 14-items assessing embarrassment related to tremor. For Score A, participants provide a simple response (disagree or agree) to each of the 14-items, the sum of which yields an initial score range = 0 to 14. Higher scores indicate greater embarrassment
Time Frame: Change from baseline to week 12
Population: The outcome was assessed in participants in the Intent to Treat (ITT) analysis population set that completed the baseline and week 12 ETEA assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | 10 Milligram (mg) JZP385 | 20 mg JZP385 | 30 mg JZP385
Number analyzed (Participants) | 98 | 99 | 95 | 97
score on a scale | -0.6 (2.84) | -0.5 (3.06) | -0.6 (3.60) | -1.2 (3.51)

11. Secondary Outcome: Change From Baseline to Week 12 on the Essential Tremor Embarrassment Assessment (ETEA) Score B as Summarized by Each Dose of JZP385 and Placebo
Description: The Essential Tremor Embarrassment Assessment (ETEA) is a participant-rated questionnaire administered by a health care provider or researcher that contains 14-items assessing embarrassment related to tremor. For Score B, participants provide a more nuanced response to each question on a 0 to 5 point Likert scale ranging from disagree (0) to agree strongly (5). The sum of the nuanced responses yields a second score (range = 0 to 70). Higher scores indicate greater embarrassment
Time Frame: Change from baseline to week 12
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | 10 Milligram (mg) JZP385 | 20 mg JZP385 | 30 mg JZP385
Number analyzed (Participants) | 98 | 99 | 95 | 97
score on a scale | -4.2 (12.87) | -3.5 (14.15) | -4.6 (14.42) | -5.6 (14.28)

ADVERSE EVENTS:
Time Frame: Up to 14 weeks
Description: A total of 420 participants were randomized to treatment. Of those 420 participants, only 416 received at least 1 dose of study intervention. Four participants did not receive any treatment. AEs were only collected in the 416 participants who received at least 1 dose of study treatment.
Arm/Group | Placebo | 10 Milligram (mg) JZP385 | 20 mg JZP385 | 30 mg JZP385
All-Cause Mortality (participants affected / at risk) | 1/104 | 0/104 | 0/103 | 0/105
Serious Adverse Events (participants affected / at risk) | 3/104 | 3/104 | 4/103 | 4/105
Other Adverse Events (participants affected / at risk) | 20/104 | 35/104 | 35/103 | 46/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=104) | 10 Milligram (mg) JZP385 (N=104) | 20 mg JZP385 (N=103) | 30 mg JZP385 (N=105)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intercostal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=104) | 10 Milligram (mg) JZP385 (N=104) | 20 mg JZP385 (N=103) | 30 mg JZP385 (N=105)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 6 (6) | 4 (5) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 6 (6) | 1 (1) | 5 (5)
Nausea (Gastrointestinal disorders) | 1 (2) | 6 (6) | 3 (3) | 4 (4)
Fatigue (General disorders) | 1 (1) | 4 (4) | 3 (3) | 7 (7)
Nasopharyngitis (Infections and infestations) | 5 (5) | 6 (6) | 0 (0) | 4 (5)
Disturbance in attention (Nervous system disorders) | 0 (0) | 2 (2) | 6 (6) | 4 (4)
Dizziness (Nervous system disorders) | 7 (9) | 11 (12) | 11 (14) | 12 (15)
Headache (Nervous system disorders) | 5 (5) | 8 (8) | 3 (3) | 5 (5)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 6 (6) | 9 (10)
Somnolence (Nervous system disorders) | 4 (4) | 2 (2) | 5 (6) | 7 (8)
Tremor (Nervous system disorders) | 2 (2) | 1 (3) | 3 (3) | 7 (7)
Anxiety (Psychiatric disorders) | 0 (0) | 6 (6) | 2 (2) | 3 (3)
Insomnia (Psychiatric disorders) | 2 (2) | 5 (5) | 3 (3) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-02-10): https://cdn.clinicaltrials.gov/large-docs/50/NCT05122650/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-31): https://cdn.clinicaltrials.gov/large-docs/50/NCT05122650/SAP_001.pdf